CLINICAL TRIAL: NCT01511341
Title: Impact of a Telenursing Service on Satisfaction and Health Outcomes of Children With Inflammatory Rheumatic Diseases and Their Family: a Crossover Trial
Brief Title: Impact of a Telenursing Service on Satisfaction and Health Outcomes of Children With Inflammatory Rheumatic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences of Western Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Réseau d'Etudes aux Confins de la Santé et du Social (RECSS)(HES-SO) (Unknown); University of Lausanne Hospitals (Other); Consultation Multisite Romande de Rhumatologie Pédiatrique (Unknown); Ligue Genevoise contre le Rhumatisme (Unknown)
Responsible Party: Principal Investigator, Anne-Sylvie Ramelet, Professor HES-S2, University of Applied Sciences of Western Switzerland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SNSF-13DPD6_132135
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Inflammatory Rheumatism
Keywords: Telenursing; Children; Chronic Illness; Nursing
MeSH Terms: conditions — Rheumatic Fever; Chronic Disease | interventions — Telenursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telenursing (Experimental)
  Interventions: Behavioral: Telenursing
- Standard practice (No Intervention): Group receive the standard practice, without telephone nursing intervention.

INTERVENTIONS:
Behavioral: Telenursing — The nurse-led intervention will consist of providing a monthly telephone call by a qualified and experienced nurse specialist in paediatric rheumatology and TN to ensure follow-up of the children and their family. The intervention will focus on providing affective support, health information, and aid to making decision.
  Arms: Telenursing

SUMMARY:
Paediatric rheumatisms represent a large group of inflammatory and non-inflammatory diseases of the locomotion system. The annual rate incidence of children diagnosed with rheumatic disease in Switzerland (canton of Vaud) is 56.8 for 100'000 children. These children experience a chronic course of the disease impacting on their quality of life and family functioning. Their medical treatment is significant and may last for life. Caring for these children involves a multidisciplinary approach. Control of the disease and management of the symptoms becomes of foremost importance to minimise disability and pain. In addition to medical care, the supporting role of nurses in the care of children with rheumatic diseases and their family aims to limit the potential for further deformity, disability, and psychological complications. In particular, they play a key role in supporting the specialist team caring for patients with rheumatism disease, recognising poor disease control and the need for changes in treatment, providing a resource to patients on treatment options and how to access additional support and advice, and identifying best practice to achieve optimal outcomes for the patients and their family. Nurses also ensure the link between medical practitioner, other health providers, and family, thus play a key role in the follow-up care of the child and its family. Follow-up of children and their family can be ensured by regular telephone consultation (telenursing) made by experienced nurse specialists in rheumatology. However, the effectiveness of telenursing remains to be proven in children with chronic rheumatic diseases. The aim of this study is, therefore, to evaluate the effect of a telephone nursing intervention on the outcomes of family and children with rheumatism chronic disease.

This randomised crossover, experimental longitudinal study will be carried out in the outpatient clinic of paediatric rheumatology of a tertiary referral hospital in canton of Vaud. The population will consist of children newly diagnosed with inflammatory rheumatologic diseases and one of their parent. The nurse-led intervention will consist of providing a monthly telephone call by a qualified and experienced nurse specialist in paediatric rheumatology and TN to ensure follow-up of the children and their family. The intervention will focus on providing affective support, health information, and aid to making decision.

ELIGIBILITY:
Inclusion Criteria:

* Children under the age of 17 years at the time of enrolment into the study
* Newly diagnosed (within 24 months from the enrolment date) with inflammatory rheumatologic diseases
* Registered as outpatient in the clinic of paediatric rheumatology
* A parent (the mother or the father or the guardian) on behalf of their children.

Exclusion Criteria:

* Children and parents who do not understand and speak French
* No access to a telephone line.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Satisfaction | 2 years
  Mixed methods, with Client Satisfaction Questionnaire (CSQ-8), and semi-structured interview

SECONDARY OUTCOMES:
Telenursing service utilisation | 2 years
  Telenursing service utilisation will be recorded in terms of number, time and duration of calls, who made the call, the nature of the call, decision made, description of the plan for action, and follow-through of the advice.
Adherence to therapeutic regimen | 2 years
  Parent Adherence Report Questionnaire (PARQ) and Child Adherence Report Questionnaire (CARQ)
Cost effectiveness | 2 years
  Cost will be descriptive in nature and be estimated by calculating the cost related to the time for the use of the service by a qualified nurse versus what the parents would have done if the service was not avalaible.
Clinical status (disease activity, QOL) | 2 years
  Juvenile Arthritis Disease Activity Score (JADAS) and Juvenile Arthritis Multidimensional Assessment Report (JAMAR)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sylvie Ramelet, PhD, Principal Investigator — Institut universitaire de formation et de recherche en soins-IUFRS
Locations (1):
- University Hospital of Vaud - Department of Pediatrics, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Ramelet AS, Fonjallaz B, Rio L, Zoni S, Ballabeni P, Rapin J, Gueniat C, Hofer M. Impact of a nurse led telephone intervention on satisfaction and health outcomes of children with inflammatory rheumatic diseases and their families: a crossover randomized clinical trial. BMC Pediatr. 2017 Jul 17;17(1):168. doi: 10.1186/s12887-017-0926-5. PMID 28716081
- [Derived] Ramelet AS, Fonjallaz B, Rapin J, Gueniat C, Hofer M. Impact of a telenursing service on satisfaction and health outcomes of children with inflammatory rheumatic diseases and their families: a crossover randomized trial study protocol. BMC Pediatr. 2014 Jun 18;14:151. doi: 10.1186/1471-2431-14-151. PMID 24939642
- See also: Swiss National Science Foundation — http://p3.snf.ch/project-132135